CLINICAL TRIAL: NCT03817814
Title: Decisions of Young Women With Breast Cancer Regarding Fertility Preservation Before Cancer Treatment and Family Building After Treatment
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-461
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Fertility Preservation; Breast Cancer
Keywords: Quality of Life; Web-based questionnaire; 18-461
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Breast Cancer: This is a cross-sectional survey of young women with breast cancer (YWBC) who received a consultation with an MSK Fertility Nurse Specialist before starting cancer treatment.
  Interventions: Behavioral: web-based questionnaire

INTERVENTIONS:
Behavioral: web-based questionnaire — Participants will complete a web-based questionnaire examining the decisions patients made about fertility preservation before and after treatment, the factors that influenced their decisions, and the ways in which patients pursue family building after treatment.

SUMMARY:
This study will help the researchers learn more about factors that affect the decisions about fertility preservation and family building made by young women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer, Stage 0-III
* Female
* 18-45 years of age at time of diagnosis
* Patients that completed their primary breast cancer treatment (surgery, chemotherapy, radiation therapy). Patients can still be on endocrine therapy, trastuzumab and/or pertuzumab therapy.
* Received education and counseling by MSK Fertility Nurse Specialist before beginning cancer treatment from 2009 through 2018

Exclusion Criteria:

* Unable to read English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with Breast Cancer Regarding Fertility Preservation before Cancer Treatment.
Study Population: This is a cross-sectional survey of YWBC who received a pre-treatment consultation with a FNS from 2009 through 2018. Participants will complete a one-time web-based questionnaire examining the decisions they made about FP before and after treatment, the factors that influenced FP decisions, and the ways in which patients pursue FB after treatment.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Patient-reported outcome questionnaire - Fertility Preservation Questionnaire | 1 year
  Number of patients reporting that fertility tools were recommended to them following their breast cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm